CLINICAL TRIAL: NCT04603638
Title: The Comparison of Analgesia Methods Used for Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dilek Hundur, Resident at Anesthesiology and Reanimation, Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/1458
Record Dates: First submitted 2020-08-09; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Analgesia; Postoperative Pain
Keywords: magnesium; morphine; scoliosis
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Scoliosis | interventions — Magnesium; N-Methylaspartate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium (Active Comparator): participations will be given intravenous magnesium.
  Interventions: Drug: Magnesium
- control (Placebo Comparator): participations will be given intravenous isotonic.
  Interventions: Drug: Isotonic

INTERVENTIONS:
Drug: Magnesium — 40 mg/kg(peroperative), 40 mg/kg (postoperative 12 h)
  Other Names: NMDA (n-metil d aspartat) blocker
  Arms: magnesium
Drug: Isotonic — 100 ml
  Other Names: Saline
  Arms: control

SUMMARY:
In this study ; Two randomized groups will be created. Iv magnesium will be given to one of the blindly designated groups. The other group will be given only isotonic. All patients will be awakened after the analgesic agents (0,1mg / kg morphine, 15mg / kg paracetamol, nsaid) are used in routine practice and will be followed up for intensive care.

The use of PCA (patient controlled analgesia) device is available in both groups.In post-operative period, magnesium infusion will be continued for 12 h. Only 100cc isotonic will be given without using magnesium to the other group. VAS (visual analog scale) score will be recorded at postoperative 30. minutes and 2,6,12,18,24 hours. In routine administration, the patient should be given 2 mg of morphine if vas>4 and the maximum dose will be increased to 10 mg.

DETAILED DESCRIPTION:
After the approval of the ethics committee for the study, in the Istanbul University Faculty of Medicine Orthopedics and Traumatology Department; There will be 3 or more posterior instrumentation operations, cobb angle of 40 degrees and above, 18-75 years old, ASA (American Society of Anesthesiologists) score 1-3, no chronic neuropathic pain and no psychiatric illness, no chronic narcotic analgesics and / or substance abuse a creatine value below 1.3 will be included.

Standard anesthesia monitoring will be performed for patients taken to the operation room. Routine anesthesia induction will be performed. In the prone position, anesthesia maintenance will be provided using the infusion of propofol and remifentanil.

Our clinic; PCA (patient-controlled analgesia) device with intravenous morphine is used routinely for postoperative analgesia.In this study ;two randomized groups will be created. It will give iv magnesium(in the intraoperative period at a dose of 40mg / kg, within 30 minutes after induction) to a blindly designated group. The other group will be given only isotonic. After in post-operative period, magnesium infusion will be continued for 12 hours (40mg / kg). Magnesium sulfate will be given in 100 cc isotonic. In the other group, only 100cc isotonic will be given without using magnesium. All patients will be awakened after the analgesic agents (0,1mg / kg morphine, 15mg / kg paracetamol, nsaid) are used in routine practice and will be followed up for intensive care.

The use of PCA device is available in both groups. vas score will be recorded postoperative 30. minutes and 2,6,12,18,24 hours. In routine administration, the patient should be given 2 mg of morphine if vas>4 and the maximum dose will be increased to 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* 18 -75 years old
* Patients with posterior instrumentation surgery of 3 or more levels under general anesthesia with a cobb angle of 40 degrees and above
* Patients who will be awakened after the surgery is completed and intensive care follow-up
* Patients with ASA classification 1-3
* Patients with creatine value <1.3 g / dl

Exclusion Criteria:

* Having a history of chronic neuropathic pain
* Having a psychiatric illness
* Patients who should not be awakened after surgery but should be followed up intubated and sedated
* Patients who cannot provide adequate cooperation for scoring
* Patients with chronic opioid use and / or substance use
* Patients with ASA classification> 3
* Patients with a creatinine value of 1.3 g / dl and higher

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-07-04 (Estimated); Study Completion 2022-02-04 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  The analgesia methods will be compared with morphine consumption
VAS score | 24 hours
  The analgesia methods will be compared with VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ilke Buget, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Jabbour HJ, Naccache NM, Jawish RJ, Abou Zeid HA, Jabbour KB, Rabbaa-Khabbaz LG, Ghanem IB, Yazbeck PH. Ketamine and magnesium association reduces morphine consumption after scoliosis surgery: prospective randomised double-blind study. Acta Anaesthesiol Scand. 2014 May;58(5):572-9. doi: 10.1111/aas.12304. Epub 2014 Mar 17. PMID 24635528